CLINICAL TRIAL: NCT02365987
Title: The Acute Effects of Interesterification of Commercially Used Fats on Postprandial Lipaemia and Satiety: a Randomised Controlled Trial. The INTER-FAT Study
Brief Title: The Acute Effects of Interesterification of Commercially Used Fats on Postprandial Lipaemia and Satiety
Acronym: INTERFAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Dr Sarah Berry, Lecturer in Nutritional Sciences, King's College London
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: BDM/14/15-26
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Healthy Men
Keywords: interesterified; postprandial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interesterified (Experimental): Interesterified blend of palm kernal and plam stearin. 50g fat.
  Interventions: Dietary Supplement: Interesterified blend of palm kernal and plam stearin
- Un-interesterified (Active Comparator): Un-interesterified blend of palm kernal and plam stearin. 50g fat.
  Interventions: Dietary Supplement: Un-interesterified blend of palm kernal and plam stearin

INTERVENTIONS:
Dietary Supplement: Interesterified blend of palm kernal and plam stearin — 50g fat provided as interesterified palm kernal and palm sterin blend in a single meal
  Other Names: Interesterified blend
  Arms: Interesterified
Dietary Supplement: Un-interesterified blend of palm kernal and plam stearin — 50g fat provided as un-interesterified palm kernal and palm sterin blend in a single meal
  Other Names: Un-interesterified blend
  Arms: Un-interesterified

SUMMARY:
The purpose of this study is to investigate whether there are differences in postprandial metabolic indices following interesterified fats used in commercial spreads versus the corresponding un-interesterified blend.

DETAILED DESCRIPTION:
Aim: The current study aims to investigate the acute effects of commercially relevant interesterified 'hardstock' versus the corresponding un-interesterified blend on postprandial lipaemia, glycaemia, insulinaemia and gut hormone responses. Due to the previously observed differences in gut hormones following interesterified palm oil and un-interesterified palm oil by our group, we will also explore acute effects of these fats on satiety and rates of gastric emptying.

Hypothesis: Interesterification of a palm kernel and palm stearin fat blend, to produce a fat with a higher proportion of palmitic acid in the middle position of the TAG (but the same fatty acid composition), will alter postprandial lipid and glucose metabolism. It is also hypothesised that differences in rates of absorption between the test fats will influence gut hormone responses and feelings of satiety.

Subjects: Participants will include 10 healthy male volunteers. In order to determine the 'typical' response to the test fats, subjects must not be affected by metabolic syndrome in any way (obesity, dyslipidemia, insulin resistance or hypertension), they must be non-smokers (since smoking influences postprandial lipaemia), and be aged between the ages of 18 and 45 years (since above this age metabolic changes may take place that may affect the way that the body digests and metabolises lipids). Male volunteers have been selected as they elicit a higher postprandial lipaemic response to a given fat load and therefore are more sensitive to dietary manipulation.

Power calculation: A sample size of 10 has 80% power to detect a difference between means of 112.74 units in area under the curve in plasma TAG with a significance level (alpha) of 0.05 (two-tailed).

Expected value:

The study will provide novel information on the acute effects of commercially relevant spreads on postprandial lipaemia and satiety. It will also explore possible mechanisms for the predicted reduced lipaemia following the interesterified fat from measurements of gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-45
2. Male
3. Healthy (free of diagnosed diseases listed in exclusion criteria)
4. Able to understand the information sheet and willing to comply with study protocol
5. Able to give informed consent

Exclusion criteria:

1. Medical history of myocardial infarction, angina, thrombosis, stroke, cancer, liver or bowel disease or diabetes
2. Body mass index < 20 kg/m2 or > 35 kg/m2
3. Plasma cholesterol ≥7.5 mmol/L
4. Plasma triacylglycerol > 3 mmol/L
5. Plasma glucose > 7 mmol/L
6. Blood pressure ≥160/100 mmHg
7. Current use of antihypertensive or lipid lowering medications
8. Alcohol intake exceeding a moderate intake (> 28 units per week)
9. Current cigarette smoker
10. ≥ 20% 10-year risk of cardiovascular disease as calculated using risk calculator
11. Ingestion of paracetamol in the preceding 24 hrs to study days

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Postprandial lipaemia (Postprandial plasma triacylglycerol concentrations) | Postprandial 4 hrs
  Postprandial plasma triacylglycerol concentrations

SECONDARY OUTCOMES:
Glycemia (Postprandial plasma glucose and insulin concentrations) | Postprandial 4 hrs
  Postprandial plasma glucose and insulin concentrations
Gut hormones (Postprandial gut peptide YY and glucose-dependent insulinotropic polypeptide concentrations) | Postprandial 4 hrs
  Postprandial gut peptide YY and glucose-dependent insulinotropic polypeptide concentrations

OTHER OUTCOMES:
Satiety (Postprandial visual analogue scales) | Postprandial 4 hrs
  Postprandial visual analogue scales
Gastric emptying (Postprandial paracetamol concentrations) | Postprandial 4 hrs
  Postprandial paracetamol concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Sarah EE Berry, BSc,MSc,PhD, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - Diabetes and Nutritional Sciences Division, School of Medicine, Kings College London, London, London
  - Diabetes and Nutritional Sciences Division, School of Medicine, Kings College London, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall WL, Iqbal S, Li H, Gray R, Berry SEE. Modulation of postprandial lipaemia by a single meal containing a commonly consumed interesterified palmitic acid-rich fat blend compared to a non-interesterified equivalent. Eur J Nutr. 2017 Dec;56(8):2487-2495. doi: 10.1007/s00394-016-1284-z. Epub 2016 Aug 10. PMID 27511058